CLINICAL TRIAL: NCT06708962
Title: Shoulder Joint Range of Motion and Subacromial Space Changes After Mulligan's Mobilization for Paraplegic Patients with Subacromial Impingement: a Randomized Controlled Trial
Brief Title: Effect of Mulligan's Mobilization on Shoulder Joint Range of Motion and Subacromial Space in Paraplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Radwa Fayek Hammam, Lecturer at Basic Science Department, MTI University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/003273
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Paraplegia, Incomplete
Keywords: Range of motion; subacromial impingement
MeSH Terms: conditions — Paraplegia; Shoulder Impingement Syndrome | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Will receive mulligan's mobilization plus corticosteroid injection for shoulder joint
  Interventions: Other: Mulligan's mobilization; Other: corticosteroid injection for rotator cuff tendinopathy
- corticosteroid injection for rotator cuff tendinopathy only (Sham Comparator): patients will receive corticosteroid injection for rotator cuff muscle only which helps in resolving inflammation at the shoulder joint
  Interventions: Other: corticosteroid injection for rotator cuff tendinopathy

INTERVENTIONS:
Other: Mulligan's mobilization — Mulligan mobilization isthe concurrent application of sustained accessory mobilization applied by a therapist and an active physiological movement to end range applied by the patient.
  Arms: Group A
Other: corticosteroid injection for rotator cuff tendinopathy — corticosteroid injection for rotator cuff helps resolving inflammation which occur for paraplegic patients from overuse of the crutches

SUMMARY:
The aim of the study is to determine the effect of mulligan's mobilization on shoulder range of motion and subacromial joint space in paraplegic patients with subacromial impingement so, thirty patients will be randomly assigned to two groups group (A) and Group (B)

DETAILED DESCRIPTION:
30 patients will be randomly assigned to two groups Group (A): will receive Mulligan's mobilization plus steroid injection for rotator cuff tendinopathy Group (B): will receive Steroid injection for rotator cuff tendinopathy only

Outcome measures will be:

* shoulder joint range of motion will be measured by laser goniometer
* Subacromial joint space will be measured by 3D ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* More than one year after traumatic spinal cord injury
* The injury is at the second thoracic level or below.
* No cognitive impairment
* Relying on manual wheelchair for main movement.

Exclusion Criteria:

* No frozen shoulder
* No subluxation

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Shoulder joint range of motion | Two months
  Shoulder joint ROM ( flexion - abduction- external and internal rotation will be measured by The laser goniometer HALO

SECONDARY OUTCOMES:
Subacromial joint space | Two months
  3D Ultrasonography enables the identification of common shoulder pathologies, and it will be utilized to assess the subacromial space as a kinematic indication of the shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Modern University for Technology and Information, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30248039/